CLINICAL TRIAL: NCT00634699
Title: Neuropathy Along the Median Nerve: Etiology of Symptoms Associated With the Carpal Tunnel Syndrome: a Preliminary Study.
Brief Title: The Treatment of Carpal Tunnel Syndrome Using Thumb Pressure Along the Median Nerve
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guy Hains Chiropractor (Other)
Responsible Party: Guy Hains DC, UQTR
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Éthic Committee, UQTR
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- One (Experimental): Ischemic Compression on Triggers Points on Muscles along the Median Nerve. Active Comparator
  Interventions: Procedure: Active Comparator, ischemic compressions

INTERVENTIONS:
Procedure: Active Comparator, ischemic compressions — Ischemic Compressions,3 times a week,5 weeks.
  Other Names: Pressure Point Therapy

SUMMARY:
The purpose of this study is to find the efficacy of treating the muscles in the inside (biceps,pronator teres) of the arm in order to eliminate the carpal tunnel syndrome .The authors hypothesise that eliminating the trigger points located in these muscles would diminish the symptoms associated with the carpal tunnel syndrome.

DETAILED DESCRIPTION:
The carpal tunnel syndrome is a common condition which should treated by surgery only when conservative approaches has been tried.In the present trial the authors intend to find the effectiveness of treating the triggers points located in the biceps muscle, the pronator teres muscle and the biceps aponeurosis on the symptoms normally associated with the carpal tunnel syndrome.

The technique used in this trial will be ischemic compression(thumb tip pressure)on the trigger points located on the previous sites.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 20 and 60 years old from the city and the surrounding Trois-Rivières with chronic carpal tunnel syndrome,
* Daily pain in the hand that lasted at least 3 months

Exclusion Criteria:

* History of upper limb or neck surgery,
* Pregnancy and systemic pathologies possibly related to carpal tunnel syndrome, such as hypothyroidism, diabetes and rheumatoid arthritis.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-09; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Pain,functional disabilities | One year

CONTACTS AND LOCATIONS:
Overall Officials: Guy Hains, DC, Principal Investigator — Université du Québec à Trois-Rivières
Locations (1):
- Guy Hains 2930 Côte Richelieu, Trois-Rivières, Quebec, Canada